CLINICAL TRIAL: NCT03901937
Title: Department of General Surgery, Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, 310016, China
Brief Title: The Effects of Parenteral ω-3 Polyunsaturated Fatty Acid on Postoperative Complications of Patients With Crohn's Disease
Acronym: ω3CD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhou, Clinical Professor, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SRRSH20180925-8
Record Dates: First submitted 2019-03-12; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Crohn Disease
Keywords: postoperative complications
MeSH Terms: conditions — Crohn Disease; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): parenteral nutrition without ω-3 polyunsaturated fatty acid
  Interventions: Drug: ω-3 polyunsaturated fatty acid; Procedure: Intestinal surgery for Crohn's Disease
- ω-3 fatty acid (Experimental): parenteral nutrition with ω-3 polyunsaturated fatty acid
  Interventions: Procedure: Intestinal surgery for Crohn's Disease

INTERVENTIONS:
Drug: ω-3 polyunsaturated fatty acid — CD patients are divided into two groups, which include with and without ω-3 polyunsaturated fatty acid-based PN (0.1-0.2g/kg/d).
  Other Names: Omegaven®10%
  Arms: Placebo
Procedure: Intestinal surgery for Crohn's Disease — Patients receive bowel resection due to complications of Crohn's Disease

SUMMARY:
This study is intended to investigate the safety and efficacy of ω-3 polyunsaturated fatty acid-based parenteral nutrition (PN) for patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis as Crohn's disease according to definition;
2. Bowel resection;
3. With parenteral nutrition at least 5 days
4. 18 years old<age<75 years old;
5. Sign the informed consent.

Exclusion Criteria:

1. Emergency surgery;
2. With severe comorbidity and/or organ (kidney,liver,or heart) dysfunction;
3. Incomplete laboratory data;
4. With parenteral nutrition before surgery;
5. Pregnant;
6. Allergy of ω-3 polyunsaturated fatty acid.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative complications | postoperative 1-30 days
  postoperative complications after surgery for Crohn's Disease according to clavien-dindo system

SECONDARY OUTCOMES:
Length of postoperative hospital stay | from surgery to discharge
  postoperative hospital stay after surgery for Crohn's Disease
Blood Concentration of IL-6 | postoperative 1, 3, and 6 day
  Blood Concentration of IL-6 after surgery
Blood Concentration of TNF-α | postoperative 1, 3, and 6 day
  Blood Concentration of TNF-α after surgery
Blood Concentration of IL-1β | postoperative 1, 3, and 6 day
  Blood Concentration of IL-1β after surgery
Blood Concentration of albumin | postoperative 1, 3, and 6 day
  Blood Concentration of albumin after surgery
Blood Concentration of C-reactive protein | postoperative 1, 3, and 6 day
  Blood Concentration of C-reactive protein after surgery
Blood White blood cell level | postoperative 1, 3, and 6 day
  Blood White blood cell level after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiujun Cai, Study Chair — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Data collection from 2019-3 to 2020-9

REFERENCES:
- [Derived] Ge X, Liu H, Wu Y, Liu W, Qi W, Ye L, Cao Q, Lian H, Bai R, Zhou W. Parenteral n-3 polyunsaturated fatty acids supplementation improves postoperative recovery for patients with Crohn's disease after bowel resection: a randomized, unblinded controlled clinical trial. Am J Clin Nutr. 2024 Apr;119(4):1027-1035. doi: 10.1016/j.ajcnut.2023.12.022. Epub 2024 Feb 19. PMID 38569774